CLINICAL TRIAL: NCT04008719
Title: Predictivity of Attention Test and Executive Functions After Stroke to Predict Depression 3 Months After Stroke.
Brief Title: ATtention Test and Executive Functions After STroke to Predict Depression.
Acronym: ATTEST-Depress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D17-P02
Record Dates: First submitted 2017-04-27; First posted 2019-07-05 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2019-07

CONDITIONS: Post-stroke Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): Assessments are made by a psychiatrist
  Interventions: Other: Thymic history; Other: Evaluation of the psychiatric disorders; Other: Cognitive evaluation

INTERVENTIONS:
Other: Thymic history — This interview concerns mainly the nature of the previous psychiatric and psychological care
Other: Evaluation of the psychiatric disorders — Mini International Neuropsychiatric Interview for the positive diagnosis of depression - under the MINI score of depression.
Other: Cognitive evaluation — They will be held consecutively to the patient's bedside interview on the same day. Some tests will be computerized, others will be in paper form.

SUMMARY:
The purpose of this study is to determine whether cognitive function evaluation (sustained attention, executive functions, working memory) during acute post-stroke is predictive of a 3 months post-stroke depression.

DETAILED DESCRIPTION:
1. Baseline visit: after neurologic stability, 14 days or less after stroke and before discharge.
2. First assessment :

   1. Neurologic data: morphologic data (MRI of the brain), stroke severity (NIHSScore), aphasia assessment (Boston Diagnostic Aphasia Examination) if NIHS verbal score ≥1, hemineglect assessment (Bells test).
   2. Personal data assessment :

   i. Socio demographic : age, gender, marital status, employment, level of education ii. Medical history: medical treatments, psychiatric and non psychiatric history.

   c. Psychiatric assessment i. Mini International Neuropsychiatric Interview - depression ii. Beck Depression Inventory iii. Clinical Global Impression iv. Standardized Assessment of Personality - Abbreviated Scale (SAPAS) v. Fageström-C vi. Alcohol Use Disorders Identification Test (AUDIT-C) d. Cognitive assessment: i. Verbal memory : Dubois's five words ii. Clock drawing test iii. D2test (computerized) iv. Verbal fluency (Cardebat) v. Working memory (digit span WAIS 3) vi. Brixton (computerized)
3. Assessment 3 months after the first assessment. Phone call and psychiatric assessment: MINI depression, Beck Depression Inventory. Barthel index and Quality of Life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Ischemic or hemorragic stroke, diagnosed with radiology : cerebral CT or MRI, 14 days or less after stroke
* Signed Consent
* Social insurance regime affiliation

Exclusion Criteria:

* Death
* No possibility of follow-up
* No French-speaker : insufficient command of French
* Deprivation of liberty : judicial or administrative decision
* D2 test assessment impossibility
* Aphasia with major disorder of the understanding (Boston <8)
* Antidepressant treatment during stroke
* Depression during stroke
* protected people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Post stroke depression | 3 months
  Whether or not a post-stroke depression occurs. occurrence of post-stroke depression assessed with Mini International Neuropsychiatric Interview (MINI), subscale depression .

SECONDARY OUTCOMES:
Post-stroke depression population characterization | 1 day
  Age, gender, marital status, occupation, level of education, laterality of stroke,and medical and psychiatric history will be collected during the inclusion interview and cognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Philip GORWOOD, MD, PhD, Study Director — CHSA
Locations (1):
- Neurology service, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided